CLINICAL TRIAL: NCT07373249
Title: The Study of Parental Toothbrushing Efficacy Assessment With Triple-Headed and Single-Headed Toothbrushes in Preschool Children With Developmental Disability: A Randomized Crossover Study
Brief Title: The Study of Parental Toothbrushing Efficacy Assessment With Triple-Headed and Single-Headed Toothbrushes in Preschool Children With Developmental Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Jantra Jitngamkusol, Principal Investigator, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MU-DT/PY-lRB 2024/ 060.2409
Record Dates: First submitted 2026-01-11; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Effectiveness of Toothbrush
Keywords: TRIPLE-HEADED TOOTHBRUSH; PLAQUE REMOVAL; DEVELOPMENTAL DISABILITY; SINGLE-HEADED TOOTHBRUSH
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triple and single headed toothbrush (Experimental): Crossover study compared effectiveness of tripled and single headed toothbrush
  Interventions: Device: Triple-headed toothbrush

INTERVENTIONS:
Device: Triple-headed toothbrush — The triple-headed toothbrush has been introduced to enhance brushing effectiveness as a design of three sides bristles, with each head capable of cleaning the buccal, lingual, and occlusal surfaces simultaneously. It is particularly suitable for individuals with limited manual skills, such as those with physical and mental handicaps, young or preschool children, especially important for caregivers when patient cooperation during brushing is limited.The round-end design is beneficial for easier brushing, reducing time, and improving cleaning efficiency, as proven in numerous studies

SUMMARY:
The Objectives

1. To evaluate the efficacy of dental plaque removal between triple-headed and single-headed toothbrushes in preschool children with developmental disabilities through parental brushing
2. To assess the parental satisfaction with triple-headed toothbrushes

DETAILED DESCRIPTION:
This study was a single-blind, randomized crossover study. 24 Parents of children with developmental disabilities (DD) were invited to participate in the study. Baseline data including demographic information, plaque index, and dmft, were collected. Participants were randomly assigned to receive their first toothbrush, either a single-head toothbrush (Berman®; soft and flat bristles for preschool children) or a triple-head toothbrush (Dr. Barman's Superbrush®; soft and flat bristles, size 0-6 years). Parents received toothbrushing instruction via a video clip according to the randomly assigned sequence of toothbrush type. Parents were then allowed to perform toothbrushing for their children. The quality of toothbrushing performance for each sextant was evaluated by the examiner using a toothbrushing performance form. Overall toothbrushing time was also recorded.

All participants were advised to use their own toothbrush during the washout period. After a four-week washout period, participants crossed over to the alternate toothbrush type, and all procedures were repeated. At the end of the study, parents completed a satisfaction questionnaire regarding the triple-headed toothbrush.

ELIGIBILITY:
Inclusion Criteria:

* Developmental disability children aged 3 to 6 years old who have full primary dentition.
* The caregivers who responsible for brushing their child's teeth that must be the same person throughout the study and able to attend both study sessions

Exclusion Criteria:

* Developmental disability children who have periodontal disease, soft tissue ulcers or gingival abscess.
* Developmental disability children who have missing tooth more than one tooth per sextant.
* Developmental disability children who have definitely negative behavior (Frankl behavior rating scale one) (89) during oral examination
* Parents of Developmental disability children who have a physical or mental disability which may influence to their brushing ability.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Dental Plaque Reduction Score Assessed by the Greene and Vermillion Plaque Index | 4 weeks per participant
  Dental plaque removal efficacy was assessed by the change in dental plaque scores measured using the Greene and Vermillion Plaque Index (score range: 0-3). Dental plaque was disclosed using Disclosing PCA 260 Liquid Solution (Curaprox, Switzerland) and evaluated on the labial/buccal and lingual/palatal surfaces of six primary teeth (teeth no. 51, 55, 65, 71, 75, and 85). Dental plaque scores were recorded immediately before and immediately after parent-performed toothbrushing using either a triple-headed toothbrush or a single-headed toothbrush, according to a randomized crossover design. The outcome measure was calculated as the difference between pre-brushing and post-brushing plaque index scores for each toothbrush type. Mean plaque score changes were compared between toothbrush types. A randomized crossover design with a four-week washout period was used to minimize carryover effects. Brushing time (in seconds) was recorded as a secondary parameter to support interpretation of pla

SECONDARY OUTCOMES:
Parental Satisfaction With the Use of a Triple-Headed Toothbrush | 4 weeks per participant
  Parental satisfaction with the triple-headed toothbrush was assessed using a self-administered satisfaction questionnaire completed after parents used the triple-headed toothbrush to brush their child's teeth.
  The questionnaire consisted of two sections. The first section collected parent demographic information, including age, sex, educational level, and relationship to the child with developmental disability. The second section assessed overall satisfaction with the triple-headed toothbrush, including ease of use, perceived effectiveness, and overall acceptance. Satisfaction responses were summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Song Hong community center for preschool mentally retarded and the Dental Department at Bangkruai Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No